CLINICAL TRIAL: NCT05708560
Title: Relationship Between Metabolic Dysfunction Associated Fatty Liver Disease and Liver Fibrosis Progression in Patients With Chronic Hepatitis B: a Multicenter Retrospective Cohort Study
Brief Title: Relationship Between MAFLD and Liver Fibrosis Progression in Patients With Chronic Hepatitis B: a Multicenter Retrospective Cohort Study
Acronym: MAFLD-HBV 1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Milan Sonneveld, dr. Milan Sonneveld, MD, PhD, Erasmus Medical Center
Other Study IDs: MEC-2021-0919
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-MAFLD, antiviral therapy
- Non-MAFLD, no antiviral therapy
- MAFLD, antiviral therapy
- MAFLD, no antiviral therapy

SUMMARY:
This multicenter retrospective study aims to study the association between the presence of MAFLD and change in liver stiffness over time in untreated and treated patients with chronic hepatitis B

DETAILED DESCRIPTION:
This project is a multicenter retrospective cohort study. All CHB patients who underwent at least 2 liver stiffness assessments with a Fibroscan device at least 6 months apart are eligible for enrolment. At baseline (defined as the first liver stiffness assessment) patients will be allocated to one of 4 groups (figure) based on use of antiviral therapy and presence of MAFLD. MAFLD is defined as presence of steatosis (based on ultrasound, histology or controlled attenuation parameter) in the presence of overweight (BMI >23 for Asians or >25 for Caucasians), diabetes mellitus, or at least 2 minor metabolic dysfunction criteria.(9) Baseline and follow-up data on biochemistry, virology, liver stiffness and clinical outcomes will be collected for all eligible patients. In case of initiation of antiviral therapy or development of MAFLD during follow-up, patients will transition to the appropriate cohort from that time-point onwards.

To ascertain the influence of the presence of MAFLD on liver stiffness progression, changes in liver stiffness will be compared within study groups (ie. cohort A vs B and cohort C vs D). To study the influence of antiviral therapy on liver stiffness progression in relation to presence of MAFLD, liver stiffness dynamics will be compared in cohort B vs cohort D (figure). The latter analysis will also be performed in the subgroup of patients with low levels of viremia (HBV DNA <2,000 IU/mL) and/or low levels of ALT (< 2 times the upper limit of normal).

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B monoinfection
* At least two liver stiffness measurements more than 6 months apart
* Availability of data on hepatic steatosis (ultrasound, controlled attenuation parameter or histology) within 1 year of baseline

Exclusion Criteria:

* antiviral therapy with drugs other than entecavir, tenofovir disoproxil fumarate or tenofovir alafenamide (for group 2 only)
* Presence of concomitant liver disease such as Wilson's disease, autoimmune hepatitis, hemochromatosis or alcohol abuse (>21 alcoholic drinks/week, female's >14/week)
* Presence of secondary causes of hepatic steatosis (medication, alcohol abuse)
* Coinfection with HCV, HIV, HEV

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis B patients
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Study the association between presence of MAFLD and change in liver stiffness over time in untreated patients with chronic hepatitis B | 12 months
Study the association between presence of MAFLD and change in liver stiffness over time in patients with chronic hepatitis B who initiate antiviral therapy | 12 months
Assess the influence of antiviral therapy on liver stiffness changes over time in CHB patients with and without MAFLD | 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Maastricht UMC+, Maastricht